CLINICAL TRIAL: NCT04741880
Title: Intravenous Lidocaine and Time to Regression of the Sensory Block After Spinal Anesthesia With Isobaric Bupivacaine in Patients Undergoing Surgery to Treat Skin and Soft Tissue Tumors of the Lower Limbs
Brief Title: Evaluation of Intravenous Lidocaine and Time to Regression of the Sensory Block After Spinal Anesthesia (ELSA Trial)
Acronym: ELSA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 40904720.3.0000.5274
Record Dates: First submitted 2021-01-28; First posted 2021-02-05 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Anesthesia; Cancer
Keywords: Spinal Anesthesia; Bupivacaine; Lidocaine; Regression of the sensory block
MeSH Terms: conditions — Neoplasms | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigators appointed for executing the protocol will not have access to the group in which the patient will be allocated. Randomization will be performed by automated system (RedCap) and at the time the investigator assigned for preparing the medication in the central pharmacy of the unit is requested to send the infusion. Only staff in the pharmacy sector will have access to the allocation group. The groups will remain masked even after closing the database and sending the data sheet for statistical analysis by the principal investigator, there will be no identification of the intervention performed in each group (lidocaine versus saline solution). After the end of the analysis, the result will be opened to finish the description of the results and develop the discussion of the findings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group L (Lidocaine) (Experimental): Lidocaine bolus 1.5 mg.kg-1 intravenous before the onset of lidocaine infusion Lidocaine 2mg.kg-1.h-1
  Interventions: Drug: Lidocaine IV
- Group S (saline solution) (Placebo Comparator): Lidocaine bolus 0.75 mg.kg-1 intravenous before the onset of saline infusion Saline solution infusion
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Lidocaine IV — Will be sent to Group L a 10 ml syringe of 2% lidocaine and 200 ml of lidocaine solution at 8mg.ml-1 (80ml of 2% lidocaine associated with 120ml 0.9% sodium chloride)
  A syringe with 10 ml of solution and a bag with 200 ml of solution indistinguishable between the groups, with the identification of the patient by label prepared specifically for the study will be prepared by the Pharmacy personal. The bag and the solution will be sealed in a waterproof and opaque envelope and sent to the Operating Theatre (OT). The envelope will be stored in the refrigerator of the sector between 3º C and 8º C until the patient is sent to the operating room, when the drugs will be sent to the operating room. At the time designated for the start of the intervention, a bolus of 0.075 ml.kg-1 of the syringe solution, followed by 0.25 ml.kg-1.h-1 in the infusion pump of the solution in the bag will be administered.
  Other Names: Lidocaine
  Arms: Group L (Lidocaine)
Drug: Saline — Group S will be sent a 10 ml syringe of 1% lidocaine and 200 ml of saline solution (0.9% sodium chloride)
  A syringe with 10 ml of solution and a bag with 200 ml of solution indistinguishable between the groups, with the identification of the patient by label prepared specifically for the study will be prepared by the Pharmacy personal. The bag and the solution will be sealed in a waterproof and opaque envelope and sent to the Operating Theatre (OT). The envelope will be stored in the refrigerator of the sector between 3º C and 8º C until the patient is sent to the operating room, when the drugs will be sent to the operating room. At the time designated for the start of the intervention, a bolus of 0.075 ml.kg-1 of the syringe solution, followed by 0.25 ml.kg-1.h-1 in the infusion pump of the solution in the bag will be administered.
  Other Names: 0.9% sodium chloride
  Arms: Group S (saline solution)

SUMMARY:
The use of intravenous lidocaine in continuous infusion in the perioperative period is associated with a reduction in postoperative pain scores, opioid use, incidence of nausea and vomiting, among other favorable outcomes. However, this therapeutic intervention has not yet been adequately evaluated by clinical trials when associated with regional anesthesia. The aim of this study is to evaluate whether the use of intravenous lidocaine in continuous infusion during spinal anesthesia with isobaric bupivacaine alters the time to regression of sensory block in patients undergoing surgical procedures for the treatment of bone and connective tissue tumor surgeries. This will be a triple-blind randomized trial. The sample size estimated was 66 patients. The study will include all patients who meet the pre-established inclusion and exclusion criteria, choose to participate, and agree with the Informed Consent Form. The main anesthetic technique will be spinal anesthesia with 13 mg of isobaric bupivacaine. Patients will be allocated in two groups in a blindly after randomization: Group S (lidocaine 0.75mg.kg-1 in bolus followed by infusion of saline solution) and Group L (lidocaine 1.5 mg.kg-1 followed by continuous infusion of lidocaine solution at 2 mg.kg-1.h-1). The primary outcome will be the time to T12 regression of the sensory block. Will also be evaluated: time to regression of the motor block, most rostral dermatome achieved by the sensory block, time to two-segment regression oh the sensory block, propofol dose in the operating room, postoperative pain score at rest, pain at movement score, quality of recovery, use of opioids in the postoperative period, nausea or vomiting, dizziness, shivering, arrhythmias, hypotension, urinary retention, and length of stay. The records will be assigned to the RedCap database. The data will be extracted without identification of the allocation groups for the R software and the groups will be revealed to the researcher after the end of the statistical analysis to write the summary of the results. The results will be submitted to scientific journals afterward.

DETAILED DESCRIPTION:
Hypotheses:

Null hypothesis

H0: The time to T12 regression of the sensory block after administration of isobaric bupivacaine is EQUAL with or without the use of intravenous lidocaine in continuous infusion.

Alternative hypothesis

H1: The time to T12 regression of the sensory block after administration of isobaric bupivacaine is DIFFERENT depending on the use or not of intravenous lidocaine in continuous infusion.

Methods

Study design

It is a randomized, controlled, triple blind clinical trial (patient, assistant team / investigator, and data collection/analysis).

Standard procedures

All patients should undergo an outpatient preoperative evaluation with an anesthesiologist. At that moment, eligibility for the study will be evaluated and the informed consent form will be presented. The preoperative form will also be completed by the investigator of the study who includes the patient of the patient.

Study participants will undergo continuous 5 leads electrocardiographic, automated noninvasive blood pressure and capnography monitoring initiated at the entrance to the operating room. Peripheral venous access will also be obtained. After certification of monitoring and venous access the patient will be positioned in lateral decubitus with the side to be performed the surgery (or the side of higher major surgical trauma in case of bilateral procedures) superiorly (e.g. surgery with right side of the body the puncture will be performed in left lateral decubitus) and then will be initiated the infusion the solutions present in the syringe and in the bag sent by the Division of Pharmacy of the hospital unit according to the protocol. Immediately after the initiation of continuous infusion of the solution the anesthesiologist will begin preparation for performing subarachnoid puncture with a Quinke needle between 22 and 27 Gauge (preferably 26 Gauge) between spaces L4-L5 and L2-L3 (preferably L3-L4) depending on the assessment of the anesthesiologist responsible for the predicted difficulty for the block and the risk of post-dural puncture headache. Conscious sedation with propofol in continuous infusion and local anesthesia with 1% lidocaine solution up to 100 mg will also be initiated. It will be administered in the subarachnoid space 13mg (2.6 ml of solution) of isobaric bupivacaine at 0.5%.

As a multimodal and antiemetic analgesia regimen, the following will be administered:

* dexamethasone 4mg in the operating room;
* ondansetron 4mg in the operating room and in case of postoperative nausea or vomiting;
* dipyrone 20mg.kg-1 every 4 hours or paracetamol 500mg every 4 hours (in case of dipyrone allergy) started before regional anesthesia and kept until discharge;
* tenoxicam 40mg in the OR and 20 mg on the first postoperative day, unless contraindicated by the assistant team;
* tramadol 50mg up to every 4 hours or morphine 4 mg up to every 10 minutes in case of pain assessed by verbal numerical scale greater than or equal to 4 (0-10) or according to evaluation of the assistant team.

After the block, evaluations of the extension of sensory and motor block will be performed at minutes 5, 10, 15 and then every 15 minutes as presented in the data collection form . The sensory block will be evaluated by pinprick sequentially from the most caudal to the most cephalic level, at the midclavicular line, on the opposite side of the surgical procedure (or on the side of minor surgical trauma in case of bilateral procedures) and will be computed as the level of blockade the point at which the patient reports sensitivity similar to reference point (homolateral shoulder) will be computed. Motor block will be initially evaluated for ankle flexion, followed by knee elevation and finally leg elevation with knees extended, and the level of motor block will be recorded according to the modified Bromage scale on the opposite side of the surgical procedure (or on the side of lower surgical trauma in case of bilateral procedures).

The patient will be released for the surgical procedure as soon as he reaches motor block evidenced by a modified Bromage scale equal to 2. During the procedure, only sensory block will be observed so that there is no interference with the surgical procedure. After the end of the procedure, each 15 minutes evaluations of sensory and motor block will be performed. Supplementary sensory and motor status evaluations may be performed in addition to the evaluations every 15 minutes at the discretion of the assistant team. After the end of the surgery. Sensory block and motor block will be evaluated concomitantly until the primary outcome (regression of sensory block up T12 dermatome), regression of motor block to modified Bromage 1 and regression of two dermatomes of the sensory block (secondary outcomes) are achieved.

The patient will be continuously evaluated in the post-anesthetic recovery room until at least the second postoperative hour and until the primary outcome. Twenty-four hours after the end of the procedure, the patient will be reevaluated at the ward, or by phone contact in case of discharge, and the study information and questionnaires will be computed as described in the data collection form.

Intervention

The bolus and infusion of the solution referring to the allocated group will be made:

* After monitoring and obtaining venous access
* Prior to the initiation of continuous propofol infusion and spinal puncture

Group L (Lidocaine):

Lidocaine bolus 1.5 mg.kg-1 intravenous before the onset of lidocaine infusion.

Lidocaine 2mg.kg-1.h-1.

Group S (saline solution):

Lidocaine bolus 0.75 mg.kg-1 intravenous before the onset of saline infusion.

Saline solution.

Group L will be sent a 20 ml syringe of 2% lidocaine and 200 ml of lidocaine solution at 8mg.ml-1 (80ml of 2% lidocaine associated with 120ml 0.9% sodium chloride) Group S will be sent a 20 ml syringe of 1% lidocaine and 200 ml of saline solution (0.9% sodium chloride)

A syringe with 20 ml of solution and a bag with 200 ml of solution indistinguishable between the groups, with the identification of the patient by label prepared specifically for the study will be prepared by the Pharmacy personal. The bag and the solution will be sealed in a waterproof and opaque envelope and sent to the Operating Theatre (OT). The envelope will be stored in the refrigerator of the sector between 3º C and 8º C until the patient is sent to the operating room, when the drugs will be sent to the operating room. At the time designated for the start of the intervention, a bolus of 0.075 ml.kg-1 of the syringe solution, followed by 0.25 ml.kg-1.h-1 in the infusion pump of the solution in the bag will be administered.

Continuous infusion of lidocaine (group L) or saline solution (group S) will be maintained until the sensory block regresses to the T12 level, until the regression of 2 dermatomes of the sensory block and until the motor block reaches the score on the modified Bromage scale 1.

The infusion will be interrupted and the masking will be broken in case of:

* severe neurological disorders (e.g. seizure, respiratory depression);
* cardiac (e.g. atrioventricular block greater than second degree, bradycardia with HR less than 40 bpm not responsive to atropine, refractory hypotension);
* other unforeseen clinical changes that pose a risk to the patient.

The infusion will be maintained until the end of anesthesia and masking in case of need for conversion to general anesthesia (e.g., insufficient block, psychomotor agitation) and the patient will be (1) censored for the outcomes related to the extension of the blockade and (2) will continue contributing to the other outcomes.

Collected variables

The variables evaluated in the study will be collected preoperatively, at the operating room, at the PACU, in the first 24 postoperative hours, and in 30 days and recorded in the RedCap database. All data collected in the study is available at the data collection sheets.

Statistical analysis

Medical records numbers and names will be included in the data collection but will not be imputed in RedCap. Therefore, the participants' data will not be revealed at the time of data extraction and analysis, preserving the anonymity of the research individuals.

The data extracted from RedCap will be analyzed in software R. The groups will be separated by intervention group, but the researcher responsible for the analysis will only have access to the groups after the end of the analysis of the results.

Continuous variables will be presented as mean and standard deviation or median and interquartile range depending on their distribution. To check the comparability between the groups and study, the basal covariates will be presented by intervention group. Bivariate statistical tests will be performed bicaudal chi-squared test, t-test, nonparametric Mann-Whitney test and log rank test depending on the characteristics of the variable. In the outcome "most rostral dermatome achieved by sensory block" each dermatome will be numbered for statistical analysis from S5 to C6 according to the following examples: S5=1, S4=2, S3=3, C8=23, C7=24 and C6=25 and will be analyzed according to its distribution. The primary outcome will be presented graphically by the Kaplan Meier curve. The value of α was set at 0.05. For the primary outcome, the p-value will be analyzed without adjustment for multiple tests. Secondary outcomes will be evaluated without adjustment for multiple comparisons because it is an exploratory analysis.

The sample size was calculation was performed with the software R, package 'WMWssp', command 'WMWssp'. Based on previous studies, the mean time for regression was estimated at 120 minutes standard deviation for sensory block regression after subarachnoid anesthesia with bupivacaine in 20 minutes. Adopting the α value of 0.05, the power of 80%, and a 10% drop out rate, the estimated sample size to demonstrate the difference of 15 minutes in the primary outcome was 66 patients (R software input: 'WMWssp(round(rnorm(1000000, 120, 20)), rnorm(1000000, 135, 20), alpha = 0.05, power = 0.8, t = 1/2, simulation = FALSE, nsim = 10^4)').

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years-old
* The American Society of Anesthesiologists (ASA) physical status classification from I to III
* To be submitted to:
* - Spinal Anesthesia
* - For surgeries performed by the Bone and Connective Tissue (TOC) service
* - Involving lower limbs and inguinal region requiring sensory block level up to the T12 dermatome (except for larger amputations and bone resections)
* - Expected duration of less than 120 minutes
* - In supine position
* That they voluntarily decide to participate in the study

Exclusion Criteria:

* Coagulation disorder that prevents the execution of the blockade:
* - International normalized ratio for prothrombin (INR) time and activity > 1.5
* - Activated partial thromboplastin time ratio (PTTa) >1.5
* - Use of enoxaparin up to 40mg/day less than 12h before the procedure
* - Use of enoxaparin above 40mg/day less than 24hours before the procedure
* - Use of oral anticoagulant or platelet aggregation inhibitors in a lower interval than recommended for spinal block
* - Other coagulation disorders that prevent spinal anesthesia
* Moderate or severe left ventricular systolic dysfunction (defined by the presence of left ventricle ejection fraction below 40%)
* Sinus bradycardia (FC < 50 beats per minute)
* Relevant cardiac conduction system disorders (e.g. atrium ventricular block greater than first-degree, Wolf-Parkinson-White syndrome)
* Clinically significant arrhythmia (e.g. atrial fibrillation)
* Body mass index (BMI) than > 35 mg.kg-1
* Previous diagnosis of liver cirrhosis
* Creatinine clearance < 30 ml/min/1.73m2 estimated by the method of the Modification of Diet in Renal Disease (MDRD) study group
* Infection at the site of lumbar puncture
* Previous spinal surgery
* Allergy to local anesthetics amino-amides
* Difficulty in communication, understanding or cognitive deficit that prevents adequate oral response to study the study forms
* Pre-existing neurological lesion in topography to be evaluated motor block
* Documented or suspected spinal or central nervous system metastasis
* Regular use of strong opioids at a dose equal or greater than 60 mg of oral morphine equivalents per day
* Desire to withdraw from the study at any time of its execution

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Time to T12 regression of the sensory block | Period: Day 0 postoperative
  Time between the injection of bupivacaine into the subarachnoid space and the regression of sensory block to T12 dermatome (in minutes)

SECONDARY OUTCOMES:
Time to motor block regression | Day 0 postoperative
  Time between the injection of bupivacaine into the subarachnoid space and the regression of motor block to the modified Bromage scale 1 (in minutes)
Most rostral dermatome achieved by the sensory block | Day 0 postoperative
  Evaluated as ordinal variable (see statistical analysis)
Time to two-segment regression of the sensory block | Day 0 postoperative
  Time between the injection of bupivacaine into the subarachnoid space and the regression of 2 dermatomes sensory block level (in minutes)
Propofol dose at the operating room | Intraoperative
  In mg
Time to the first opioid rescue | Intraoperative
  In mg
Postoperative pain score at rest | Admission to the PACU, 2 postoperative hours, 24 postoperative hours, and worse in the first 24 postoperative hours measurements
  Verbal numerical scale between 0 and 10, being 0 = "no pain" and 10 = "worst pain imaginable"
Pain score at movement | 24 postoperative hours
  Verbal numerical scale between 0 and 10, being 0 = "no pain" and 10 = "worst pain imaginable"
Quality of recovery in 24 hours | 24 postoperative hours
  Quality of recovery measured by the "40-item quality-of-recovery questionnaire" (QoR-40)
Need for opioid analgesics (binary) | Between 0 and 6 postoperative hours, between 6 and 24 postoperative hours, and between 0 and 24 postoperative hours
  YES/NO
Need for opioid analgesics (continuous) | between 0 and 6 postoperative hours, between 6 and 24 postoperative hours, and between 0 and 24 postoperative hours
  In oral morphine equivalents (in mg)
Nausea or vomiting | Between 0 and 6 postoperative hours, between 6 and 24 postoperative hours, and between 0 and 24 postoperative hours
  Presence of nausea or vomiting reported by the patient - YES/NO
Dizziness | From intraoperative to 24 postoperative hours
  Report of dizziness by patient - YES/NO
Bradycardia | At the operating room (OR) and admission to the PACU up to 24 postoperative hours
  Heart rate below 50 beats per minute (YES/NO)
Other arrhythmias | At the OR and admission to the PACU up to 24 postoperative hours
  Heart rhythm change except sinus bradycardia and sinus tachycardia (YES/NO)
Hypotension | At the OR, between 0 and 6 postoperative hours, between 6 and 24 postoperative hours, and between 0 and 24 postoperative hours
  MAP < 65mmHg or presence of compatible symptoms (such as nausea, vomiting or cognitive impairments)
Urinary retention | Between 0 and 24 postoperative hours
  Voiding difficulty that requires bladder catheterization for relief by the assistant team
Length of stay | Through study completion, an average of 30 days
  Time between the end of the operation and administrative discharge in days

CONTACTS AND LOCATIONS:
Overall Officials: Bruno LC Araujo, MSc, EDAIC, Principal Investigator — Department of Anesthesiology, Hospital do Câncer II, Instituto Nacional do Câncer
Locations (1):
- Hospital de Câncer II, INCA, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller RD. Miller's Anesthesia. 7th ed. Phyladelphia: Churchill Livingstone/Elsevier; 2010.
- [Background] Imbelloni LE, Moreira AD, Gaspar FC, Gouveia MA, Cordeiro JA. Assessment of the densities of local anesthetics and their combination with adjuvants: an experimental study. Rev Bras Anestesiol. 2009 Mar-Apr;59(2):154-65. doi: 10.1590/s0034-70942009000200003. English, Portuguese. PMID 19488527
- [Background] Lui AC, Polis TZ, Cicutti NJ. Densities of cerebrospinal fluid and spinal anaesthetic solutions in surgical patients at body temperature. Can J Anaesth. 1998 Apr;45(4):297-303. doi: 10.1007/BF03012018. PMID 9597201
- [Background] Beloeil H. Opioid-free anesthesia. Best Pract Res Clin Anaesthesiol. 2019 Sep;33(3):353-360. doi: 10.1016/j.bpa.2019.09.002. Epub 2019 Sep 26. PMID 31785720
- [Background] Blaudszun G, Lysakowski C, Elia N, Tramer MR. Effect of perioperative systemic alpha2 agonists on postoperative morphine consumption and pain intensity: systematic review and meta-analysis of randomized controlled trials. Anesthesiology. 2012 Jun;116(6):1312-22. doi: 10.1097/ALN.0b013e31825681cb. PMID 22546966
- [Background] Gelineau AM, King MR, Ladha KS, Burns SM, Houle T, Anderson TA. Intraoperative Esmolol as an Adjunct for Perioperative Opioid and Postoperative Pain Reduction: A Systematic Review, Meta-analysis, and Meta-regression. Anesth Analg. 2018 Mar;126(3):1035-1049. doi: 10.1213/ANE.0000000000002469. PMID 29028742
- [Background] Ng KT, Yap JLL, Izham IN, Teoh WY, Kwok PE, Koh WJ. The effect of intravenous magnesium on postoperative morphine consumption in noncardiac surgery: A systematic review and meta-analysis with trial sequential analysis. Eur J Anaesthesiol. 2020 Mar;37(3):212-223. doi: 10.1097/EJA.0000000000001164. PMID 31977626
- [Background] Wang X, Lin C, Lan L, Liu J. Perioperative intravenous S-ketamine for acute postoperative pain in adults: A systematic review and meta-analysis. J Clin Anesth. 2021 Feb;68:110071. doi: 10.1016/j.jclinane.2020.110071. Epub 2020 Oct 26. PMID 33007645
- [Background] Weibel S, Jokinen J, Pace NL, Schnabel A, Hollmann MW, Hahnenkamp K, Eberhart LH, Poepping DM, Afshari A, Kranke P. Efficacy and safety of intravenous lidocaine for postoperative analgesia and recovery after surgery: a systematic review with trial sequential analysis. Br J Anaesth. 2016 Jun;116(6):770-83. doi: 10.1093/bja/aew101. PMID 27199310
- [Background] Hermanns H, Hollmann MW, Stevens MF, Lirk P, Brandenburger T, Piegeler T, Werdehausen R. Molecular mechanisms of action of systemic lidocaine in acute and chronic pain: a narrative review. Br J Anaesth. 2019 Sep;123(3):335-349. doi: 10.1016/j.bja.2019.06.014. Epub 2019 Jul 11. PMID 31303268
- [Background] Dunn LK, Durieux ME. Perioperative Use of Intravenous Lidocaine. Anesthesiology. 2017 Apr;126(4):729-737. doi: 10.1097/ALN.0000000000001527. No abstract available. PMID 28114177
- [Background] Ghimire A, Subedi A, Bhattarai B, Sah BP. The effect of intraoperative lidocaine infusion on opioid consumption and pain after totally extraperitoneal laparoscopic inguinal hernioplasty: a randomized controlled trial. BMC Anesthesiol. 2020 Jun 3;20(1):137. doi: 10.1186/s12871-020-01054-2. PMID 32493276
- [Background] Farag E, Ghobrial M, Sessler DI, Dalton JE, Liu J, Lee JH, Zaky S, Benzel E, Bingaman W, Kurz A. Effect of perioperative intravenous lidocaine administration on pain, opioid consumption, and quality of life after complex spine surgery. Anesthesiology. 2013 Oct;119(4):932-40. doi: 10.1097/ALN.0b013e318297d4a5. PMID 23681143
- [Background] Choi GJ, Kang H, Ahn EJ, Oh JI, Baek CW, Jung YH, Kim JY. Clinical Efficacy of Intravenous Lidocaine for Thyroidectomy: A Prospective, Randomized, Double-Blind, Placebo-Controlled Trial. World J Surg. 2016 Dec;40(12):2941-2947. doi: 10.1007/s00268-016-3619-6. PMID 27379388
- [Background] Beaussier M, Delbos A, Maurice-Szamburski A, Ecoffey C, Mercadal L. Perioperative Use of Intravenous Lidocaine. Drugs. 2018 Aug;78(12):1229-1246. doi: 10.1007/s40265-018-0955-x. PMID 30117019
- [Background] Gustafsson UO, Scott MJ, Schwenk W, Demartines N, Roulin D, Francis N, McNaught CE, Macfie J, Liberman AS, Soop M, Hill A, Kennedy RH, Lobo DN, Fearon K, Ljungqvist O; Enhanced Recovery After Surgery (ERAS) Society, for Perioperative Care; European Society for Clinical Nutrition and Metabolism (ESPEN); International Association for Surgical Metabolism and Nutrition (IASMEN). Guidelines for perioperative care in elective colonic surgery: Enhanced Recovery After Surgery (ERAS((R))) Society recommendations. World J Surg. 2013 Feb;37(2):259-84. doi: 10.1007/s00268-012-1772-0. No abstract available. PMID 23052794
- [Background] Melloul E, Lassen K, Roulin D, Grass F, Perinel J, Adham M, Wellge EB, Kunzler F, Besselink MG, Asbun H, Scott MJ, Dejong CHC, Vrochides D, Aloia T, Izbicki JR, Demartines N. Guidelines for Perioperative Care for Pancreatoduodenectomy: Enhanced Recovery After Surgery (ERAS) Recommendations 2019. World J Surg. 2020 Jul;44(7):2056-2084. doi: 10.1007/s00268-020-05462-w. PMID 32161987
- [Background] Nygren J, Thacker J, Carli F, Fearon KC, Norderval S, Lobo DN, Ljungqvist O, Soop M, Ramirez J; Enhanced Recovery After Surgery (ERAS) Society, for Perioperative Care; European Society for Clinical Nutrition and Metabolism (ESPEN); International Association for Surgical Metabolism and Nutrition (IASMEN). Guidelines for perioperative care in elective rectal/pelvic surgery: Enhanced Recovery After Surgery (ERAS((R))) Society recommendations. World J Surg. 2013 Feb;37(2):285-305. doi: 10.1007/s00268-012-1787-6. No abstract available. PMID 23052796
- [Background] Khezri MB, Rajabi M, Yaghoobi S, Barikani A. Effect of intravenous lignocaine infusion on bispectral index during spinal anaesthesia for caesarean section: A prospective randomised double-blind study. Indian J Anaesth. 2020 May;64(5):369-374. doi: 10.4103/ija.IJA_424_19. Epub 2020 May 1. PMID 32724244
- [Background] Levey AS, Coresh J, Greene T, Stevens LA, Zhang YL, Hendriksen S, Kusek JW, Van Lente F; Chronic Kidney Disease Epidemiology Collaboration. Using standardized serum creatinine values in the modification of diet in renal disease study equation for estimating glomerular filtration rate. Ann Intern Med. 2006 Aug 15;145(4):247-54. doi: 10.7326/0003-4819-145-4-200608150-00004. PMID 16908915
- [Background] Park SK, Lee JH, Yoo S, Kim WH, Lim YJ, Bahk JH, Kim JT. Comparison of bupivacaine plus intrathecal fentanyl and bupivacaine alone for spinal anesthesia with intravenous dexmedetomidine sedation: a randomized, double-blind, noninferiority trial. Reg Anesth Pain Med. 2019 Apr;44(4):459-465. doi: 10.1136/rapm-2018-100084. Epub 2019 Jan 23. PMID 30679336
- [Background] Verret M, Lauzier F, Zarychanski R, Perron C, Savard X, Pinard AM, Leblanc G, Cossi MJ, Neveu X, Turgeon AF; Canadian Perioperative Anesthesia Clinical Trials (PACT) Group. Perioperative Use of Gabapentinoids for the Management of Postoperative Acute Pain: A Systematic Review and Meta-analysis. Anesthesiology. 2020 Aug;133(2):265-279. doi: 10.1097/ALN.0000000000003428. PMID 32667154